CLINICAL TRIAL: NCT03060486
Title: A New Approach for Controlling Hemostasis During Canal Treatment: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Riccardo Pace (Other)
Responsible Party: Sponsor-Investigator, Dr Riccardo Pace, Principal Investigator, Azienda Ospedaliero-Universitaria Careggi
Organization: Azienda Ospedaliero-Universitaria Careggi (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: endo1-2016
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Results first posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Blood Contamination of Root Canal During Endodontic Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HYBENX® (Experimental): 1 cc of mixture of hydroxybenzenesulfonic acid (37%) and hydroxymethoxybenzene acids (23%), sulfuric acid (28%), and water (12%) for 20 sec
  Interventions: Device: HYBENX®

INTERVENTIONS:
Device: HYBENX® — The mixture was then introduced inside the root canal using the pre-dosed syringe for 20 seconds with a sterile paper point with and up and down movement.
  Finally, the canal was rinsed with sterile saline water using a syringe with a side-vented 30 G needle.

SUMMARY:
Blood contamination, such as apical microleakage, of root canal during preparation can be a major problem in endodontics. The purpose of this investigation was to evaluate the hemostatic properties of sulfonic/sulfuric acid solution used during root canal therapy in teeth with irreversible pulpitis.

DETAILED DESCRIPTION:
A new device (HYBENX®) has been developed with the purpose of destroying dental biofilm. The material contains a concentrated aqueous mixture of hydroxybenzenesulfonic acid (37%) and hydroxymethoxybenzene acids (23%), sulfuric acid (28%), and water (12%).

The investigators planned a clinical and microbiological study using the decontaminant device in order to destroy the dental biofilm of root canals in cases of irreversible pulpitis. The ability of the decontaminant device to immediately stop bleeding during canal instrumentation was found out accidentally during the procedures of this still unpublished trial.

Due to this fact, the investigators were interested in evaluating the coagulation property of the material. Therefore, the aim of this prospective study is to describe a new approach to obtain hemostasis during root canal therapy using a sulfonic/sulfuric acid solution.

A total of 15 teeth with irreversible and acute pulpitis were included in the study. After manual and mechanical instrumentation of the root canal, a sterile paper point was introduced in the canal, and a first score was given based on the blood quantity.

The solution was used to irrigate the bleeding root canal; then a second sterile paper point was introduced, and the same score was assessed. The null hypothesis was that there is no difference in root canal bleeding before and after the use of the solution (⎧=0)

ELIGIBILITY:
Inclusion Criteria:

* tooth affected by irreversible pulpitis, single-rooted teeth associated with healthy periodontium, physiologic sulcus depth (<3 mm), and absence of bleeding on probing of the involved teeth.

Exclusion Criteria:

* patients with systemic diseases using anticoagulants, antibiotics, or anti-inflammatory therapies in the last 30 days, patients with allergy to sulfur in any form, and pregnancy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-17 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Teeth
Groups:
- HYBENX®: 1 cc of mixture of hydroxybenzenesulfonic acid (37%) and hydroxymethoxybenzene acids (23%), sulfuric acid (28%), and water (12%) for 20 sec
  HYBENX®: The mixture was then introduced inside the root canal using the pre-dosed syringe for 20 seconds with a sterile paper point with and up and down movement.
  Finally, the canal was rinsed with sterile saline water using a syringe with a side-vented 30 G needle.
Period: Overall Study
Arm/Group | HYBENX®
Started | 15; 15 Teeth
Completed | 15; 15 Teeth
Not Completed | 0; 0 Teeth

BASELINE CHARACTERISTICS:
Arm/Group | HYBENX®
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Root Canal Bleeding Score
Description: After the root canal, shaping was performed, and a first sterile paper point was introduced in the root canal, up to the working length, to detect blood presence.
  The root canal bleeding score (RCBS) was given as follows:
  * 0: no blood detected
  * 1: blood detected in the apical third of the root canal
  * 2: blood detected both in the apical and the middle thirds of the root canal
  * 3: blood detected in the whole root canal. After the use of the material a second sterile paper point was introduced in the root canal, up to the working length, to detect the presence of blood and an RCBS was assessed according the previous criteria
Time Frame: 20 sec - before and after use
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: teeth
Arm/Group | HYBENX®
Number analyzed (Participants) | 15
Number analyzed (teeth) | 15
score on a scale
  Before use | 2.33 (0.724)
  After use | 0.13 (0.352)
Statistical Analysis 1: Comparison: HYBENX®; Test type: Other; p < .0001, Wilcoxon signed-rank test; Signed Rank Score Difference = -60

ADVERSE EVENTS:
Arm/Group | HYBENX®
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes